CLINICAL TRIAL: NCT01144936
Title: A Phase 1b, Randomized, Double-Blind, Placebo-Controlled, Multiple-Dose Study of VX-985 in Subjects With Genotype 1 Chronic Hepatitis C
Brief Title: Study of VX-985 in Subjects With Chronic Hepatitis C
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Lisa Mahnke, Vertex Pharmaceuticals Incorporated
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX09-985-101
Record Dates: First submitted 2010-06-14; First posted 2010-06-16 (Estimated); Last update posted 2011-03-09 (Estimated); Status verified 2011-03

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Panel 1: VX-985 Dose 1 (Experimental)
  Interventions: Drug: VX-985 or matching placebo
- Panel 2: VX-985 Dose 2 (Experimental)
  Interventions: Drug: VX-985 or matching placebo
- Panel 3: VX-985 Dose 3 (Experimental)
  Interventions: Drug: VX-985 or matching placebo

INTERVENTIONS:
Drug: VX-985 or matching placebo — low dose
  Arms: Panel 1: VX-985 Dose 1
Drug: VX-985 or matching placebo — high dose
  Arms: Panel 2: VX-985 Dose 2
Drug: VX-985 or matching placebo — dose TBD
  Arms: Panel 3: VX-985 Dose 3

SUMMARY:
The purpose of this study it to evaluate the safety and tolerability of VX-985 in HCV subjects. This study will also evaluate the antiviral activity and pharmacokinetic profile of VX-985.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are male or females of non-childbearing potential aged 18 to 64 years(inclusive) with a body mass index (BMI) between 18 and 32 (kg/m2)
* Certain subjects must agree to use acceptable contraceptive methods as specified in protocol
* Subjects who are treatment naïve and are infected with genotype 1 chronic hepatitis C
* Subjects must be in good health and have normal laboratory values as judged by investigator
* Subjects must not have clinically significant abnormal results for physical examination

Exclusion Criteria:

* Subjects must not have received approved or experimental HCV therapy
* Subjects must not have evidence of hepatic decompensation: history of ascites, hepatic encephalopathy, or bleeding esophageal varices
* Subjects must not have any known history of other cause of significant liver disease including hepatitis B, drug or alcohol-related cirrhosis, etc
* Subjects must not be diagnosed with or have suspected hepatocellular carcinoma
* Subjects must not have histologic evidence of hepatic cirrhosis on any liver biopsy or test capable of detecting cirrhosis within the past 2 years
* Subjects with a known history or other evidence of severe retinopathy or clinically significant ophthalmological disorder
* Subjects must not have a history of any illness that might confound the results of the study or pose an additional risk in administering study drug(s) to the subject e.g. history of cardiovascular or central nervous system disease, ongoing psychiatric disorder, poorly controlled diabetes, etc
* Subject must not have taken any of the prohibited medications within the specified time before study start or take certain medications (including herbal supplements) during the study
* Subjects must not have a history of drug or alcohol abuse or addiction within 6 months before the start of dosing, or test positive for alcohol or drugs of abuse
* Subjects must not have donated or had a significant loss of blood within 56 days of the start of dosing, or donated more than 1 unit of plasma within 7 days before the start of dosing
* Subjects must not consume excessive amounts of caffeine
* Subjects must not have participated in a clinical study involving administration of either an investigational or a marketed drug within 2 months
* Subjects who are female and have a positive pregnancy test and/or who are considered to be of childbearing potential or are nursing.
* Subjects that have a female partner who is pregnant, nursing, or planning to become pregnant during the study or shortly after the study

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Estimated)
Dates: Start 2010-06; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability (vital signs, 12-lead electrocardiograms, physical examinations, laboratory assessments, and adverse events) | 10-13 days

SECONDARY OUTCOMES:
Plasma pharmacokinetic parameters of VX-985 | 10-13 days
HCV RNA levels | 5-7 months

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Mahnke, MD, PhD, Study Director — Vertex Pharmaceuticals Incorporated
Locations (3):
- United States (3):
  - Kansas, Overland Park, Kansas
  - Maryland, Baltimore, Maryland
  - Washington, Tacoma, Washington